CLINICAL TRIAL: NCT02712918
Title: An Evaluation of Brief Behavioral Activation Treatment for Depression With Moderate to Severely Depressed Inpatients - A Small Randomized Controlled Trial
Brief Title: Brief Behavioral Activation Treatment for Depression With Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Martin Myhre, Learning Disability Nurse/MSc Behavior Analysis, Lovisenberg Diakonale Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BATD_16674
Record Dates: First submitted 2015-03-09; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: Depression; Inpatient; Acute; Brief Behavioral Activation Treatment for Depression
MeSH Terms: conditions — Depression | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Behavioral Activation Treatment for Depression (Experimental): Behavioral treatment of depression. The study utilized the revised version of the Brief Behavioral Activation Treatment for Depression (BATD) protocol from 2011. The treatment was added to treatment as usual. Up to 10 sessions were administered.
  Interventions: Behavioral: Brief Behavioral Activation Treatment for Depression
- Standard care (Placebo Comparator): Standard CARE (SC) at the inpatient unit. Mandatory: Therapeutic conversations with psychiatrist, psychologist or M.D, milieu therapy. Optional: Psychosomatic physiotherapy, therapeutic groups, psychopharmacological treatment.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Brief Behavioral Activation Treatment for Depression — Behavioral treatment of depression which focuses on increasing the Level of positive reinforcement through systematic and goal directed activation of behavior. Goal and values are assessed and used to determine target behaviors.
  Arms: Brief Behavioral Activation Treatment for Depression
Other: Standard Care — Treatment as usual at the ward
  Arms: Standard care

SUMMARY:
The purpose of the current study was to examine Brief Behavioral Activation Treatment for Depressions (BATD) effectiveness, credibility, and acceptability with moderate to severly depressed inpatients. The study is a systematic replication of a randomized controlled trail from 2003, that provided initial support for BATD With inpatients. The current study compared BATD to Treatment as Usual in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe depression (BDI-II > 28 Points).
* Admission length of at least 3 days
* Evaluated to benefit from depression treatment by unit psychiatrist.

Exclusion Criteria:

* Current psychotic disorder
* Previously diagnosis with psychotic disorder (including Bipolar disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change of Beck's Depression Inventory-II from baseline | Change from baseline (second day of admission) to discharge from the ward (maximum 21 days, expected average of 10 days).

SECONDARY OUTCOMES:
Credibility and Expectancies Questionnaire | Second day of admission. After first sessions of BATD.
  Only BATD group
Treatment Evaluation Inventory - Short Form | Prior to discharge from the ward (maximum 21 days, expected average of 10 days)..
  Only BATD group

REFERENCES:
- [Background] Lejuez CW, Hopko DR, Hopko SD. A brief behavioral activation treatment for depression. Treatment manual. Behav Modif. 2001 Apr;25(2):255-86. doi: 10.1177/0145445501252005. PMID 11317637
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Result] Hopko DR, Lejuez CW, LePage JP, Hopko SD, McNeil DW. A brief behavioral activation treatment for depression. A randomized pilot trial within an inpatient psychiatric hospital. Behav Modif. 2003 Sep;27(4):458-69. doi: 10.1177/0145445503255489. PMID 12971122